CLINICAL TRIAL: NCT04975932
Title: Efficacy and Safety of Transarterial Chemoembolization in Combination With Immune Checkpoint Inhibitors for Hepatocellular Carcinoma: a Real-world Study
Brief Title: Efficacy and Safety of TACE in Combination With ICIs for HCC: a Real-world Study
Acronym: CHANCE001
Status: Completed | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: TACE-ICIs-RWS
Record Dates: First submitted 2021-07-02; First posted 2021-07-26 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; transarterial chemoembolization; immune checkpoint iInhibitors; real-world study
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: TACE+ICIs: TACE: cTACE (conventional TACE) or dTACE (drug-eluting beads TACE); ICIs: atezolizumab, pembrolizumab, nivolumab, camrelizumab, tislelizumab, sintilimab or other ICIs
  Interventions: Other: TACE+ICIs
- Control group: TACE: TACE: cTACE (conventional TACE) or dTACE (drug-eluting beads TACE);
  Interventions: Procedure: TACE

INTERVENTIONS:
Other: TACE+ICIs — TACE plus ICIs ( with or without molecular targeted therapies)
  Groups: Study group: TACE+ICIs
Procedure: TACE — TACE without combination of ICIs ( with or without molecular targeted therapies)
  Groups: Control group: TACE

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of transarterial chemoembolization (TACE) in combination with immune checkpoint inhibitors (ICIs) in patients with hepatocellular carcinoma (HCC) .

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) can induce immunogenic cell death and tumor-specific immune response which results in the release of tumor antigens and transform "cold" tumors with lacking immune effector cells into "hot" tumors with immune effector cells infiltration. This provides a theoretical basis for TACE combined with immune checkpoint inhibitors (ICIs) in hepatocellular carcinoma (HCC) patients. The purpose of this study is to evaluate the safety and efficacy of TACE in combination with ICIs in patients with HCC. This real-world study also explores the optimal combined treatment and outcome of HCC patients for providing further information for clinical practice and trials.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with HCC by radiology, histology, or cytology;
2. patients who underwent TACE combined with ICIs therapies ( with or without molecular targeted therapies) were included in the study group. For patients in the study group, ICIs therapies were received before the TACE or within 2 months after TACE and at least one cycle of immunotherapy has been received;
3. during the same period, patients who underwent TACE without the combination of ICIs therapies ( with or without molecular targeted therapies) were included into the control group;
4. patients who underwent TACE combined with ICIs therapies and molecular targeted therapies, molecular targeted therapies must be performed simultaneously with TACE or immunotherapy.

Exclusion Criteria:

1. exceeding the time interval of the combination therapy defined above;
2. missing follow-up data;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC who are candidates for TACE combined with ICIs therapies under real-world practice conditions.
Sampling Method: Non-Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival(PFS) | up to approximately 1 years
  The PFS is defined as the time from the initiation of any combination treatment to progression according to mRECIST or death from any cause. When pseudoprogression is suspected by investigator, tumor response will be re-assessed per iRECIST to confirm (also applicable for secondary endpoint of efficacy).

SECONDARY OUTCOMES:
Overall survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death from any cause.
Time to Progression(TTP) | up to approximately 1 years
  The TTP is defined as the time from the initiation of any combination treatment to progression according to mRECIST. When pseudoprogression is suspected by investigator, tumor response will be re-assessed per iRECIST to confirm.
Objective response rate(ORR) | 6-8 week after TACE
  The ORR is defined as the proportion of patients with a documented complete response or partial response per mRECIST.
Disease control rate(DCR) | 6-8 week after TACE
  The DCR is defined as the proportion of patients with a documented complete response, partial response, or stable disease according to mRECIST.
Adverse event(AE) | baseline to end of study (approximately 2 years)
  Number and degree of the AEs according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Gao-Jun Teng, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu HD, Li HL, Huang MS, Yang WZ, Yin GW, Zhong BY, Sun JH, Jin ZC, Chen JJ, Ge NJ, Ding WB, Li WH, Huang JH, Mu W, Gu SZ, Li JP, Zhao H, Wen SW, Lei YM, Song YS, Yuan CW, Wang WD, Huang M, Zhao W, Wu JB, Wang S, Zhu X, Han JJ, Ren WX, Lu ZM, Xing WG, Fan Y, Lin HL, Zhang ZS, Xu GH, Hu WH, Tu Q, Su HY, Zheng CS, Chen Y, Zhao XY, Fang ZT, Wang Q, Zhao JW, Xu AB, Xu J, Wu QH, Niu HZ, Wang J, Dai F, Feng DP, Li QD, Shi RS, Li JR, Yang G, Shi HB, Ji JS, Liu YE, Cai Z, Yang P, Zhao Y, Zhu XL, Lu LG, Teng GJ; CHANCE001 Investigators. Transarterial chemoembolization with PD-(L)1 inhibitors plus molecular targeted therapies for hepatocellular carcinoma (CHANCE001). Signal Transduct Target Ther. 2023 Feb 8;8(1):58. doi: 10.1038/s41392-022-01235-0. PMID 36750721
- [Result] Jin ZC, Zhong BY, Chen JJ, Zhu HD, Sun JH, Yin GW, Ge NJ, Luo B, Ding WB, Li WH, Chen L, Wang YQ, Zhu XL, Yang WZ, Li HL, Teng GJ; CHANCE Investigators. Real-world efficacy and safety of TACE plus camrelizumab and apatinib in patients with HCC (CHANCE2211): a propensity score matching study. Eur Radiol. 2023 Dec;33(12):8669-8681. doi: 10.1007/s00330-023-09754-2. Epub 2023 Jun 27. PMID 37368105